CLINICAL TRIAL: NCT02011815
Title: A Prospective Study of Exploring Possible Biological Linkage Between Circadian Disruption and Cancer Progression
Brief Title: Exploring Biological Linkage Between Circadian Disruption and Cancer Progression
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BreastCA_circa_mech
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2018-04

CONDITIONS: Breast Neoplasms
Keywords: Breast neoplasms; Circadian rhythm; sleep; survival; distress; anxiety; depression; quality of life; actigraph; fatigue
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum Saliva Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast cancer: Diagnosed breast cancer patients who are getting chemotherapy for the first time.

SUMMARY:
The purpose of this study is to explore the possible association between the circadian disruption and cancer progression.

DETAILED DESCRIPTION:
The biological markers that are assumed to bridge this association are measured and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70
* Breast cancer patients who are getting chemotherapy for the first time in life
* Patients are either having stage 4 cancer or starting neoadjuvant chemotherapy.
* Patient have signed on the informed consent, and well understood the objective and procedure of this study

Exclusion Criteria:

* Patients already have received chemotherapy
* Patient had another cancer (except thyroid cancer) within 5 years
* Patient with severe medical condition
* Patient had taken psychiatric medication more than 1 month in life
* Patient worked the night shift for more than 1 month in 6 months

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University (Tertiary) hospital, oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2013-11-10 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 3 years (and more) after recruitment
  The data progression-free survival will be done by reviewing patients' medical record.

SECONDARY OUTCOMES:
Circadian disruption | Baseline, after 1 month, after 6 month, after 12 month
  Morningness-Eveningness Questionnaire and Munich Chronotype Questionnaire will be used during assessment.
Objective sleep cycle measures | Baseline, after 1 month, after 6 month, after 12 month
  The assessment will be performed by using actigraph and sleep diary.
Physiological measures | Baseline, after 1 month, after 6 month, after 12 month
  The measures include blood pressure, body temperature, skin conductance, breathing pattern, and Electroencephalography.
Sleep quality measures | Baseline, after 1 month, after 6 month, after 12 month
  The measurements will be performed using Epworth sleepiness scale, Pittsburgh Sleep Quality Index, and Insomnia Severity Index.
Quality of Life measure | Baseline, after 1 month, after 6 month, after 12 month
  The measurement will be performed using M.D. Anderson Symptom Inventory.
Cancer related Fatigue | Baseline, after 1 month, after 6 month, after 12 month
  Fatigue severity scale will be used during the assessment.
Distress related measure | Baseline, after 1 month, after 6 month, after 12 month
  Hospital Anxiety and Depression Scale will be used during the assessment.
Posttraumatic Stress-related symptom measure | Baseline, after 1 month, after 6 month, after 12 month
  Impact of Event Scale-revised will be used to categorize and quantify Posttraumatic stress-related symptom in cancer patients.
Menopausal symptom measure | Baseline, after 1 month, after 6 month, after 12 month
  Menopause Rating Scale will be used during the assessment.
Personality measure | Baseline
  Temperament and Character Inventory will be used to examine the personality factor in each participant.
Genetic polymorphism | Baseline
  Variable Number Tandem Repeat and Single Nucleotide Polymorphism of circadian-rhythm related genes will be examined.
Epigenetic Change | Baseline
  The methylation specific Polymerase Chain Reaction technique will be used to explore methylation patterns in circadian clock gene or in a global gene level.
Cortisol level | Baseline
  Salivary cortisol level will be measured multiple times at baseline.
Melatonin | Baseline
  Salivary or Urine melatonin level will be measured.
Inflammatory markers | Baseline
  The various inflammation markers will be measured from blood sample.
Overall survival | 3 years (and more) after recruitment
  The data progression-free survival will be done by reviewing patients' medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Jin Hahm, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

REFERENCES:
- See also: study site webpage — http://www.snuh.org/
- See also: Institutional Review Board — https://cris.snuh.org/ncris/